CLINICAL TRIAL: NCT07142824
Title: Comparison Between Burn Dressing Using Tilapia-Fish Skin Versus Regular Dressing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Osama Mohmoud Elsherief, Resident, Department of Plastic Surgery, Faculty of Medicine, Sohag University, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med--25-8-6MS
Record Dates: First submitted 2025-08-13; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- burn dressing using Tilapia-Fish Skin (Active Comparator): we use tilapia fish skin as a healing dressing in burn patients
  Interventions: Procedure: burn dressing using Tilapia-Fish Skin
- burn dressing using regular dressing (Active Comparator): we use regular dressing in burn patients
  Interventions: Procedure: burn dressing using regular dressing

INTERVENTIONS:
Procedure: burn dressing using Tilapia-Fish Skin — we use tilapia fish skin as a healing dressing in burn patients
  Arms: burn dressing using Tilapia-Fish Skin
Procedure: burn dressing using regular dressing — we use regular dressing in burn patients
  Arms: burn dressing using regular dressing

SUMMARY:
The aim of this study is to evaluate the use of tilapia fish skin as a healing dressing in burn patients and its clinical outcome and compare it with regular dressing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with second or third-degree burns.

Exclusion Criteria:

* Patients with first-degree burns.
* Patients with burn injuries complicated by sepsis.
* Patients who received prior wound healing agents.
* Elderly patients or those with chronic diseases such as diabetes mellitus.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Effect of burn dressing using Tilapia-Fish Skin versus regular dressing on wound healing | 3 weeks after regular dressing
  Time of healing process

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] Dhivya S, Padma VV, Santhini E. Wound dressings - a review. Biomedicine (Taipei). 2015 Dec;5(4):22. doi: 10.7603/s40681-015-0022-9. Epub 2015 Nov 28. PMID 26615539
- [Background] Hu Z, Yang P, Zhou C, Li S, Hong P. Marine Collagen Peptides from the Skin of Nile Tilapia (Oreochromis niloticus): Characterization and Wound Healing Evaluation. Mar Drugs. 2017 Mar 30;15(4):102. doi: 10.3390/md15040102. PMID 28358307
- [Background] Ibrahim A, Soliman M, Kotb S, Ali MM. Evaluation of fish skin as a biological dressing for metacarpal wounds in donkeys. BMC Vet Res. 2020 Dec 3;16(1):472. doi: 10.1186/s12917-020-02693-w. PMID 33272259